CLINICAL TRIAL: NCT00148109
Title: Phase II Trial of Cetuximab in Patients With Metastatic and/or Locally Advanced Soft Tissue and Bony Sarcomas
Brief Title: Trial of Cetuximab in Patients With Metastatic and/or Locally Advanced Soft Tissue and Bony Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2004-078; Legacy IRB #2005-0072 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2011-09-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Sarcoma
Keywords: Unresectable/metastatic high grade soft tissue bony sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGFR positive (Active Comparator): The EGFR positive group will be conducted in a 2-stage minimax trial design to determine the rate of four-month progression free survival in this patient population treated with cetuximab
  Interventions: Drug: Cetuximab
- EGFR Negative (Active Comparator): The EGFR negative group will help us explore the possibility of benefit of cetuximab in a patient whose tumor does not express or minimally expresses EGFR. If benefit in progression-free survival or in another surrogate such as tumor response or a molecular event is seen in this group it would provide rationale to study this group further in subsequent trials
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — The initial dose of cetuximab is 400 mg/m2 intravenously administered over 120 minutes, followed by weekly infusions at 250 mg/m2 IV over 60 minutes.
  Arms: EGFR positive
Drug: Cetuximab — Cetuximab 400 mg/m2 over 120 min IV initial does followed by weekly Cetuximab 250 mg/m2 over 60 min
  Arms: EGFR Negative

SUMMARY:
The purpose of this study is to explore how this cancer is affected by a new medication, cetuximab. Cetuximab is directed towards a protein called EGFR (epidermal growth factor receptor), that is found in some types of cancer. Studies have shown that this drug can be beneficial in patients with colon cancer and has been approved by the US Food and Drug Administration (FDA) for this purpose. The researchers are conducting a study to see if it is beneficial in patients with sarcoma.

DETAILED DESCRIPTION:
Sarcomas are mesenchymal malignancies that arise in the connective tissue throughout the body and afflict approximately 11,000 people in the United States yearly. Sarcomas are heterogeneous with well over 50 subtypes described. The peak incidence is subtype-specific with certain sarcomas seen in children and young adults while other subtypes peak in late middle-age, causing significant morbidity and mortality in young patients and productive adults.

The precise etiology for most sarcomas remains unknown. External radiation therapy is an established risk factor. Other risk factors include occupational exposures to certain chemicals, lymphedema, and hereditary conditions such as neurofibromatosis and Li-Fraumeni syndrome. Many sarcomas are associated with specific somatic genetic alterations. For example, some specific subtypes are associated with gene translocations causing aberrant fusion proteins including Ewing sarcoma (EWS-FLI-1), synovial sarcoma (SSX-SYT), alveolar rhabdomyosarcoma (PAX3-FHKR), and myxoid liposarcomas (TLS-CHOP). These singular molecular alterations imply that some sarcomas are cytogenetically simple and may be more appropriate substrates for therapy targeted to a single molecular pathway.

Sarcomas are commonly present as an asymptomatic mass or with local symptoms in an extremity or the retroperitoneum. Although tumor size, location, and histologic subtype have been implicated as prognostic factors in sarcomas, histologic grade remains the most important factor. Tumor grade is based on the degree of cellularity, differentiation, pleomorphism, necrosis, and the number of mitoses. Approximately 50-60% of patients with high grade soft tissue sarcoma will eventually have metastatic disease, as compared to 5-10% of patients with low grade disease.

Sarcomas spread hematogenously with the most common site of spread being the lung, followed by liver, bone, and brain. About 50% of patients with sarcoma eventually expire due to locally advanced or metastatic disease with a median survival of 8-12 months.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, patients must fulfill all of the following criteria:

1. Patients must have the ability to give informed consent and have signed an approved informed consent form.
2. Patients must have a pathologic diagnosis of soft tissue sarcoma or bony sarcoma.
3. Patients with tumor tissue available for assessment of EGFR status performed by immunohistochemistry (IHC).
4. Patients with Zubrod performance status 0-2.
5. Patients must be 16 years of age or older.
6. Patients, 16 years or older, must either be not of child bearing potential or have a negative pregnancy test within 7 days of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
7. If patients are childbearing or have child-fathering potential, they must use barrier contraception during intercourse while being treated on this study.
8. Bone marrow function: absolute neutrophil count (ANC) 1,000/ul; platelets 75,000/l.
9. Renal function: creatinine 2.0 x institutional upper limit of normal (ULN).
10. Hepatic function: bilirubin 2.5 x ULN; AST 5.0 x ULN.
11. Patients must have received at least one systemic chemotherapy treatment or else refuse to be treated with cytotoxic therapy.
12. Twenty-eight days or more should have elapsed since the patient has received any prior systemic therapy.
13. Patients must have documented symptomatic or radiologic progression to their preceding therapy.
14. For patients treated with prior radiation, 21 days or more should have elapsed since the administration of the last fraction of radiation therapy and patients must have recovered from all associated toxicities.
15. Patients must have measurable disease. The measurable lesion should be outside previously irradiated fields or have documented progression at least 6 weeks after completion of radiation.

Exclusion Criteria:

Any of the following criteria will make the patient ineligible to participate in this study:

1. Acute hepatitis or known HIV.
2. Active or uncontrolled infection.
3. Significant history of uncontrolled cardiac disease i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
4. Prior therapy which specifically and directly targets the EGFR pathway.
5. Prior severe infusion reaction to a monoclonal antibody.
6. Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).
7. Other active systemic malignancy within the past year.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-06; Primary Completion 2008-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Chugh, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 subjects were recruited between June of 2005 and June of 2008 in the Comprehensive Cancer Center outpatient Oncology Clinics at the University of Michigan Health Systems
Pre-assignment Details: Potential participants who appeared to meet study criteria were approached with a brief discussion of the study. If interested, a more in - depth detail discussion of the risks and benefits of potentially participating in the study took place with the subject as well as any family members that may have been present.
Groups:
- Epidermal Growth Factor Receptor Negative: Sarcoma does not express Epidermal growth factor receptor. Patients received cetuximab 400 mg per meter squared IV followed by 250 mg per meter squared weekly
- Epidermal Growth Factor Receptor Positive: Sarcoma expresses Epidermal growth factor receptor. Patients received cetuximab 400 mg per meter squared IV followed by 250 mg per meter squared weekly
Period: Overall Study
Arm/Group | Epidermal Growth Factor Receptor Negative | Epidermal Growth Factor Receptor Positive
Started | 15 | 21
Completed | 3 | 1
Not Completed | 12 | 20
Not completed — Lack of Efficacy | 10 | 18
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidermal Growth Factor Receptor Negative | Epidermal Growth Factor Receptor Positive | Total
Number analyzed (Participants) | 15 | 21 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 1 | 4 | 5
Age Continuous [Median (Full Range); unit: years] | 49 (2) [23 to 77] | 54 (2) [29 to 78] | 54 (2) [23 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 5 | 14 | 19
Region of Enrollment [Number; unit: participants]
  United States | 15 | 21 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Sarcoma Who Are Tumor Progression Free and Alive at Four Months From Start of Treatment With Single-agent Cetuximab.
Description: Time of cetuximab administration to clinically documented progression of disease or death assessed for four months after starting cetuximab therapy
Time Frame: 4 months
Population: per protocol all patients that received drug were evaluated for the primary endpoint
Measure: Number; unit: participants
Groups:
- Epidermal Growth Factor Receptor Negative: Tumor did not express epidermal growth factor receptor
- Epidermal Growth Factor Receptor Positive: Tumor did express epidermal growth factor receptor
Arm/Group | Epidermal Growth Factor Receptor Negative | Epidermal Growth Factor Receptor Positive
Number analyzed (Participants) | 15 | 21
participants | 3 | 1
Statistical Analysis 1: Comparison: Epidermal Growth Factor Receptor Negative vs Epidermal Growth Factor Receptor Positive; Estimate a 4 month progression-free survival rate for each group; Test type: Superiority or Other; p < 0.05, Fisher Exact

2. Secondary Outcome: Progression Free Survival.
Description: Time of cetuximab administration to clinically documented progression of disease or death assessed for four months
Time Frame: survival
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Epidermal Growth Factor Receptor Negative | Epidermal Growth Factor Receptor Positive
Number analyzed (Participants) | 15 | 21
months | 1.8 [0.8 to 2.5] | 1.7 [1.6 to 1.8]

3. Secondary Outcome: Overall Survival
Description: Time of cetuximab administration to clinically documented death assessed for four months
Time Frame: months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Epidermal Growth Factor Receptor Negative | Epidermal Growth Factor Receptor Positive
Number analyzed (Participants) | 15 | 21
months | 15.7 [7.7 to 25.3] | 7.7 [4.2 to 10.7]

ADVERSE EVENTS:
Arm/Group | Epidermal Growth Factor Receptor Negative | Epidermal Growth Factor Receptor Positive
Serious Adverse Events (participants affected / at risk) | 9/15 | 10/21
Other Adverse Events (participants affected / at risk) | 10/15 | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidermal Growth Factor Receptor Negative (N=15) | Epidermal Growth Factor Receptor Positive (N=21)
spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) — unrelated to treatment. Related to tumor progession of underlying disease
Acute Neurological Symptoms (Nervous system disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Bacterial meningitis (Infections and infestations) | 0 (0) | 1 (1)
Chest Pressure and Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower GI Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
intestinal ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Vascular disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Vertigo (Vascular disorders) | 0 (0) | 0 (0)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidermal Growth Factor Receptor Negative (N=15) | Epidermal Growth Factor Receptor Positive (N=21)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 11 (11) — diffuse erythemitus rash
Nausea/vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Fatigue (General disorders) | 6 (6) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
infusion reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) — allergic reaction to infusion

LIMITATIONS AND CAVEATS:
accrual to EGFR + cohort suspended after first step for lack of efficacy of cetuximab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No